CLINICAL TRIAL: NCT02656251
Title: Efficacy of Two Clorhexidine Formulations to Control the Initial Subgingival Biofilm Formation
Brief Title: Efficacy of Two Chlorhexidine Solutions to Control the Initial Subgingival Biofilm Formation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Patricia Weidlich, Doctor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: URio Grande
Record Dates: First submitted 2015-11-18; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Dental Plaque
Keywords: biofilms; cross over trial; chlorhexidine
MeSH Terms: conditions — Dental Plaque | interventions — Ethanol; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.12% Clorhexidine with alcohol (Active Comparator): 0.12% Clorhexidine with alcohol, 15ml every 12 hour for 4 days
  Interventions: Drug: 0.12% Clorhexidine with alcohol; Drug: placebo; Drug: 0.12% Clorhexidine without alcohol
- 0.12% Clorhexidine without alcohol (Experimental): 0.12% Clorhexidine without alcohol, 15ml every 12 hour for 4 days
  Interventions: Drug: 0.12% Clorhexidine with alcohol; Drug: placebo; Drug: 0.12% Clorhexidine without alcohol
- control (Placebo Comparator): placebo 15ml every 12 hour for 4 days
  Interventions: Drug: 0.12% Clorhexidine with alcohol; Drug: placebo; Drug: 0.12% Clorhexidine without alcohol

INTERVENTIONS:
Drug: 0.12% Clorhexidine with alcohol — Use of 0.12% Clorhexidine with alcohol every 12 hours for 04 days
  Other Names: Periogard; No plak
Drug: placebo — Use of placebo every 12 hours for 04 days
Drug: 0.12% Clorhexidine without alcohol — Use of 0.12% Clorhexidine without alcohol, every 12 hours for 04 days
  Other Names: Periogard

SUMMARY:
The aim of the study is to compare the effect of a suspension containing chlorhexidine and alcohol and another one containing clorhexidine with no alcohol in dynamic of the subgingival biofilm formation versus a Placebo suspension. The initial subgingival biofilm formation will be evaluated by means of Plaque Free Zone (PFZ).

DETAILED DESCRIPTION:
This is a double blind, cross over, randomized clinical trial. 35 volunteers will stop mechanical supragingival biofilm removal measures for 96h following a complete scaling and polishing of the tooth surfaces. During this period they will be asked to rinse for a minute a Solution containing chlorhexidine and alcohol or a solution with chlorhexidine alcohol-free or placebo. Every 24h the presence of deposits will be registered with special attention to the presence of a plaque free zone between the apical border of the deposits and the gingival margin. Absence of deposits is scored 0, presence of deposits and plaque free zone =1 and presence of deposits and absence of plaque free zone =2 (MALISKA, A. N. et al. Measuring early plaque formation clinically. Oral health preventive dentistry, v. 4, p. 273-278, 2006). The prevalence of scores and the rate of changes from scores 0 and 1 into 2 will be evaluated for significance. Sample size was calculated taking the results from the study o MALISKA, AN (2006) as reference.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 years;
* non-smokers;
* have good general health;
* present at least 20 natural teeth in the mouth, including the incisors, canines and premolars without restorations, crowns, gingival recession, anatomic defects, gingivitis e/or periodontitis.

Exclusion Criteria:

* • positive history of using antibiotic e/or anti-inflammatory drugs in the month previous to the initial consultation;

  * positive history of allergies at using Triclosan;
  * pregnant or lactating patients;
  * patients in use of fixed orthodontic appliance.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of two clorhexidine formulations to Control the Initial Subgingival Biofilm Formation assessed by the plaque free zone index. | 24hours
  The presence of scores 0, 1 or 2 of the index "Plaque Free Zone" will be recorded at baseline and at each 24 hours, during a period of 96 hours (4 days).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Weidlich, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil